CLINICAL TRIAL: NCT01834976
Title: Observational Study of Cardiac Biomarker During Perioperative Management in Pediatric Heart Disease
Brief Title: Cardiac Biomarker in Pediatric Heart Disease
Status: Completed | Type: Observational
Sponsor: Okayama University (Other)
Responsible Party: Principal Investigator, Tomoyuki Kanazawa, Pediatric cardiac surgery investigators, Okayama University
Other Study IDs: pchd biomarker in okayama
Record Dates: First submitted 2013-04-15; First posted 2013-04-18 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Congenital Heart Disease
Keywords: cardiac biomarker; congenital heart disease; surgery
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum,urine

SUMMARY:
The purpose of this study is to investigate cardiac biomarker during perioperative management in pediatric cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* children who receive surgery for congenital heart disease
* require cardiopulmonary bypass for surgery
* under 18 years old

Exclusion Criteria:

* simple congenital heart disease (atrial septal defect, ventricle septal defect, patent ductus arteriosus)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric patients who receive surgery for congenital heart disease under 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2012-11; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
serious adverse events | one month

CONTACTS AND LOCATIONS:
Locations (1):
- Okayama University Hospital, Okayama, Okayama-ken, Japan